CLINICAL TRIAL: NCT01358890
Title: Effect of Low-Carbohydrate or Restricted-Calories Diet on Body Weight
Brief Title: Low-Carbohydrate Diet Intervention on Body Weight
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Chinese Academy of Sciences (Other Government)
Collaborators: Harvard School of Public Health (HSPH) (Other)
Responsible Party: Principal Investigator, Xu Lin, Principal Investigator, Chinese Academy of Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 30930081/C150502-LC
Record Dates: First submitted 2011-05-23; First posted 2011-05-24 (Estimated); Last update posted 2012-02-28 (Estimated); Status verified 2012-02

CONDITIONS: Over Weight; Obesity
Keywords: over weight; obesity
MeSH Terms: conditions — Obesity | interventions — Diet, Carbohydrate-Restricted

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- B (Experimental): Subjects will be supplied with low carbohydrate diet for 12 weeks.
  Interventions: Other: low carbohydrate diet
- A (Experimental): Subjects will be supplied with calories restricted diet for 12 weeks
  Interventions: Other: Calories restricted diet

INTERVENTIONS:
Other: low carbohydrate diet — Dietary carbohydrate diet was restricted to 20 gram/day within the first week, then increase gradually to 120 gram/day
  Arms: B
Other: Calories restricted diet — Total energy intake is restricted to 1200 kcal/day for women. Energy from carbohydrate, protein and fat will be kept to approximate 55%, 20% and 25%, respectively. Moreover, saturated fat and dietary cholesterol are restricted to at most 10% energy and 300 mg/day, respectively
  Arms: A

SUMMARY:
* The primary aim of this study is to determine the adherence of low- carbohydrate among Chinese.
* Then compare the effect of low-carbohydrate and traditional Chinese but restricted-calories diet on weight loss and metabolic traits.

DETAILED DESCRIPTION:
Obesity is a well established risk factor for type 2 diabetes mellitus, hypertension, dyslipidemia and cardiovascular disease. Along with rapid nutritional and lifestyle transition featured as increased energy dense diet intake and reduced physical activity, the prevalence of obesity has reached epidemic level and affected more than 70 million Chinese adults nowadays. Previous studies suggested that low-carbohydrate diet was an effective and safe way to lose weight and had potential benefit on lipids profiles. However, it is still unknown whether this diet can be feasible to control the epidemic of obesity and its related metabolic diseases among Chinese, whose carbohydrate consumption contribute approximately 55% of total energy intake.

Therefore, the aim of this pilot study is to investigate the adherence and effectiveness of two weight-loss diets among Chinese. This will be a randomized, controlled clinical trial. A total of 50 overweight or obese nurse assistants will be randomly assigned to receive a low-carbohydrate diet or a traditional high-carbohydrate Chinese but restricted-calories diet for 12 weeks. The adherence of study protocol and effects of the two diets on body weight, waist circumference, body fat, fasting glucose and lipid profile will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* overweight/obese (BMI ≥24 kg/m2)

Exclusion Criteria:

* Pregnancy or lactation;
* Serum creatinine and blood urea nitrogen level beyond the clinical reference value;
* alanine aminotransferase and aspartate aminotransferase beyond the reference levels;
* Gastrointestinal problems that would prevent them from complying with the specified feeding conditions;
* Received gastrointestinal surgery (except for appendicitis or hernia);
* Severer CVD;
* Active cancer;
* Mental diseases, epilepsia or using anti-depression drugs;
* Participating in other scientific studies within 3 months before the study.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-05; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
weight | 12 weeks

SECONDARY OUTCOMES:
body fat mass | 12 weeks
waist circumference | 12 weeks
body mass index | 12 weeks
fast glucose | 12 weeks
total cholesterol | 12 weeks
triglyceride | 12 weeks
LDL-C | 12 weeks
HDL-C | 12 weeks
blood pressure | 12 weeks
urinary ketone | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Xu Lin, PhD, Principal Investigator — Institute for Nutritional Sciecnes, Chinese Acadamy of Sciences
Locations (1):
- Institute for Nutritional Sciences, Chinese Academy of Sciences, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Ma Y, Sun Y, Sun L, Liu X, Zeng R, Lin X, Li Y. Effects of gut microbiota and fatty acid metabolism on dyslipidemia following weight-loss diets in women: Results from a randomized controlled trial. Clin Nutr. 2021 Nov;40(11):5511-5520. doi: 10.1016/j.clnu.2021.09.021. Epub 2021 Sep 23. PMID 34656033